CLINICAL TRIAL: NCT05030025
Title: Single-Dose Fasting and Fed Pilot BE Study in Healthy Males and Females Not of Childbearing Potential
Brief Title: Abacavir, Dolutegravir and Lamivudine Dispersible Tablets (60 mg/5 mg/30 mg)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABDL-TBP-1001
Record Dates: First submitted 2021-07-28; First posted 2021-09-01 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — abacavir; dolutegravir; Lamivudine; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: Single-dose, randomized, two-period, two-treatment, two-group, crossover study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): single-dose pharmacokinetics will be characterized in twenty-four (24) healthy, adult males and females not of childbearing potential under fasting conditions.
  Interventions: Combination Product: abacavir, dolutegravir and lamivudine dispersible tablets; Combination Product: Triumeq Dispersible Tablets 5 mg GSK1349572 [Dolutegravir]/ 60 mg Abacavir/ 30 mg Lamivudine
- Group 2 (Experimental): single-dose pharmacokinetics will be characterized in twenty-four (24) healthy, adult males and females not of childbearing potential under fed conditions.
  Interventions: Combination Product: abacavir, dolutegravir and lamivudine dispersible tablets; Combination Product: Triumeq Dispersible Tablets 5 mg GSK1349572 [Dolutegravir]/ 60 mg Abacavir/ 30 mg Lamivudine

INTERVENTIONS:
Combination Product: abacavir, dolutegravir and lamivudine dispersible tablets — Abacavir, Dolutegravir and Lamivudine Dispersible Tablets, 60 mg/5 mg/30 mg Dose: 60 mg/5 mg/30 mg (1 x 60 mg/5 mg/30 mg)
  Other Names: fixed combination
Combination Product: Triumeq Dispersible Tablets 5 mg GSK1349572 [Dolutegravir]/ 60 mg Abacavir/ 30 mg Lamivudine — Triumeq Dispersible Tablets 5 mg GSK1349572 [Dolutegravir]/ 60 mg Abacavir/ 30 mg Lamivudine Dose: 60 mg/5 mg/30 mg (1 x 60 mg/5 mg/30 mg)
  Other Names: Triumeq

SUMMARY:
The rationale for this study is to evaluate and understand the variability of a generic alternative of abacavir, dolutegravir and lamivudine dispersible tablets for PEPFAR submission to aide in the development of pivotal studies.

DETAILED DESCRIPTION:
This study is to investigate the bioequivalence of Mylan's abacavir, dolutegravir and lamivudine dispersible tablets, 60 mg/5 mg/30 mg to ViiV's Triumeq Dispersible Tablets (5 mg GSK1349572 [dolutegravir]/ 60 mg abacavir/ 30 mg lamivudine) following administration of a single, oral 60 mg/5 mg/30 mg (1 x 60 mg/5 mg/30 mg) dose of Mylan's abacavir, dolutegravir and lamivudine dispersible tablets or ViiV's Triumeq Dispersible Tablets administered under fasting and fed conditions.

Adverse events will be monitored to ensure the safety and well-being of the healthy volunteers.

ELIGIBILITY:
Inclusion Criteria - Subject candidates must fulfill all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

* 18 to 55 years old.
* Males and/or females not of child-bearing potential.
* Each subject is required to weigh at least 50 kg (110 lbs) for men and 48 kg (106 lbs) for women and have a Body Mass Index (BMI) value less than or equal to 30.0 kg/m2 but greater than or equal to 19.0 kg/m2.
* Adequate venous access in both arms.
* Only non-tobacco/non-nicotine subjects.
* Able to understand and sign the written Informed Consent Form.
* Willing to follow the protocol requirements and comply with protocol restrictions.
* All subjects should be judged by the Principal Investigator or Medical Sub- Investigator as normal and healthy during a pre-study medical evaluation performed within 28 days of the initial dose of study medication.

Exclusion Criteria - Subject candidates must not be enrolled in the study if subject meet any of the following criteria:

* Institutionalized subjects.
* Social Habits, Medications and Diseases will be evaluated.
* Use of certain foods and processed candies, gums food/drinks that contain sugar alcohols.
* Liver function tests (ALT, AST and total bilirubin).
* Subjects who are positive for the HLA-B*5701 allele.
* Subjects having Modified Patient Health Questionnaire (PHQ)-12 questionnaire score > 4.
* Subject has a creatinine clearance < 90 mL/min, as determined by the Cockroft-Gault equation.
* Any reason which, in the opinion of the Principal Investigator or Medical Sub- Investigator, would prevent the subject from safely participating in the study.
* Intolerance to venipuncture.
* Donation or loss of blood or plasma.
* Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* Allergy or hypersensitivity to abacavir, dolutegravir, lamivudine, other related products, or any inactive ingredients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 2 weeks
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 2 weeks
  Plasma concentration-time curve from zero to the time of the last measurable time point t
Area under the plasma concentration versus time curve (AUC)0-∞ | 2 weeks
  Area under the plasma concentration-time curve from zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Lawrence, Ph.D., Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Altasciences, Montreal, Quebec, Canada